CLINICAL TRIAL: NCT01104090
Title: Initial Experience With Storz C-MAC Video Intubation System
Acronym: C-MAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Davide Cattano, Associate Professor - Anesthesiology, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: HSC-MS-09-0161
Record Dates: First submitted 2010-04-13; First posted 2010-04-15 (Estimated); Results first posted 2021-11-01 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Intubation; Difficult
Keywords: C-MAC; direct laryngoscopy; indirect laryngoscopy; to determine the safety and efficacy of the C-MAC

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- C-MAC direct laryngoscopy, then C-MAC indirect laryngoscopy (Experimental): Patients assigned to this arm will be intubated using C-MAC with direct laryngoscopy first and then using C-MAC with indirect laryngoscopy.
  Interventions: Device: C-MAC direct laryngoscopy; Device: C-MAC Indirect laryngoscopy
- C-MAC indirect laryngoscopy, then C-MAC direct laryngoscopy (Experimental): Patients assigned to this arm will be intubated using C-MAC with indirect laryngoscopy first and then using C_MAC with direct laryngoscopy.
  Interventions: Device: C-MAC direct laryngoscopy; Device: C-MAC Indirect laryngoscopy

INTERVENTIONS:
Device: C-MAC direct laryngoscopy — Patients will be intubated using C-MAC with direct laryngoscopy.
Device: C-MAC Indirect laryngoscopy — Patients will be intubated using C-MAC with indirect laryngoscopy.

SUMMARY:
The purpose of this study is to determine the safety and efficacy of the C-MAC (Karl Storz Endoscopy, Inc., Tuttlingen, Germany) video intubation system guided intubation techniques.

We hypothesize that the C-MAC video laryngoscope is safe and efficacious in terms of successful endotracheal intubation. The C-MAC may be a safe and suitable alternative device for routine and difficult laryngoscopy and tracheal intubation. This is the first study to investigate the performance of C-MAC in clinical practice.

DETAILED DESCRIPTION:
Since the introduction of the laryngoscope into clinical anesthesia practice, innovators have attempted to improve upon and perfect the design of the laryngoscope blade. The goal of these innovations has been to improve visualization of laryngeal structures and increase the likelihood of successful tracheal intubation.

It is estimated that endotracheal intubation is performed on some 8 million patients per year in the United States. Of these endotracheal intubations, approximately 80% are performed by direct laryngoscopy with transoral placement of the endotracheal tube (ET) into the trachea. The incidence of unsuspected difficult intubation is estimated to be higher at approximately 3%. One factor that contributes to difficult intubation is poor visualization of the airway.

Video laryngoscopes are a relatively new edition to the armamentarium of airway devices available to the airway manager. Although these instruments are more expensive than traditional direct laryngoscopes, they offer several advantages that may justify their expense. While many clinicians may espouse the routine use of video laryngoscopy, most providers advocate its use for anticipated difficult situations, or as "plan B" after failed intubation by direct laryngoscopy (DL).

The video laryngoscopes have been shown to provide superior views to traditional laryngoscopy in normal and difficult intubation situations.3-6 Video intubation techniques, by allowing tracheal intubation monitoring, improve the safety of the procedure and increase intubation success. In contrast, using conventional laryngoscopy, anesthesiologists have only a "keyhole" view of the airway structures; a view that may be further obscured during attempts to pass the ET tube.

The C-MAC video laryngoscope is the latest edition to the pool of video laryngoscopes. C-MAC is a further development of the V-MAC (Karl Storz Endoscopy, Inc., Tuttlingen, Germany) video laryngoscope. The C-MAC became commercially available in US in March 2009 and at this time; there are no studies available regarding its use in clinical practice.

The device consists of a laryngoscope handle and Macintosh blade that have been modified to provide a video image of airway structures on a screen, which can be conveniently located directly in front of the anesthesiologist. A micro video module based on CMOS image sensor technology is contained in the modified handle and an image/light bundle is introduced into the standard blade. Because of its design, this is the video laryngoscope system which can be used to perform either a direct or indirect laryngoscopy.

A. General Study Design-

The study will include a total of 50 patients. All patients will be intubated using conventional endotracheal tube preferably without any alternative aid.

In the operating room, standard monitoring devices will be applied including a pulse oximeter, 3 lead (at least), ECG and blood pressure cuff; the latter could be invasive or non-invasive depending on the nature of the surgery. Baseline measures of BP, pulse, oxygen saturation, and CO2, will be made. The time will be noted before any sedation or anesthesia is administered. Vital signs will be recorded every minute from the time that induction of anesthesia is begun until five minutes after the patient has been intubated, and then at five-minute intervals thereafter for fifteen minutes.

General anesthesia will be induced by bolus administration of propofol (2-3 mg/kg) and fentanyl (1-2 mcg/kg), and maintained with an inhalational agent. Rocuronium (0.6 mg/kg) will be administered, after face mask ventilabilty being checked, to provide muscle relaxation and a mixture of sevoflurane or isoflurane and nitrous oxide (per anesthesiologist choice) will be utilized for maintenance of anesthesia once the ability to mask ventilate is confirmed. The lungs will be mechanically ventilated with a semi-closed circle system to maintain an end-tidal CO2 near 35 mmHg. Patients' lungs will be ventilated via an anesthesia mask for five minutes with 100% oxygen until the patient is completely relaxed.

All investigators, residents and attendings, will be trained based on manufacturer recommendations, and each resident will perform at least 3 intubations with C-MAC video laryngoscope prior to enlisting any patients for the study. Intubations will be performed by 2nd and 3rd year (CA-2 and CA-3) residents. The resident will perform direct laryngoscopy utilizing C-MAC followed by the video laryngoscopy or vice versa. In an effort to prevent bias, a computer-generated list will be prepared to help randomize the order of execution between direct laryngoscopy and indirect video laryngoscopy; intubations will be performed during the second method used. The resident will first take a direct look at the larynx without manipulating the scope. Then, the resident will take a video-assisted look (or vice versa). Subsequently, the operator will compare the direct view with the video-assisted view, then intubate. He/she will record an observation of the laryngeal aperture for both based on the Cormack-Lehane Scale and a percentage of glottic opening score (POGO Score). External neck pressure may be applied by an assistant in an attempt to improve exposure of the larynx. The anesthesiologist's assessment of the optimal view obtained by these maneuvers will be recorded.

To clarify, residents will have only one attempt opportunity each for direct laryngoscopy and in-direct video assisted laryngoscopy. If, after the first unsuccessful attempt, the attending anesthesiologist will take one more attempt respectively for the direct and in-direct views. Between laryngoscopy attempts, the intubator will achieve easy patient ventilation before the next attempt is made. The number of attempts (maximum 4 total) measured as either the reinsertion of the blade or endotracheal tube) and the intubation time (time the laryngoscope blade enters the mouth until 1st capnograph breath) will also be recorded. If unsuccessful, the direct laryngoscopy/ flexible fibreoptic laryngoscopy will be performed to intubate the trachea. If more than 4 attempts (two maximum for each type of laryngoscopy) were needed or if the anesthesiologist discontinued use of the video laryngoscope, the case will be deemed a failure. The subjective level of difficulty (from 0 = Extremely Easy to 5 = Extremely Difficult) in the performance of intubation will also be recorded.

There is a plan to do the second phase of the study. This will include a total of 50 patients with anticipated difficult airway (limited mouth opening, restricted neck movement, Mallampati 4, thyromental distance < 6 cm, BMI ≥ 40 kg/m2). All patients will be adult surgical candidates aged 18-80 years, ASA I- III, presenting for elective surgery who require general endotracheal anesthesia. We hypothesize that the C-MAC may be a safer and suitable alternative device for both routine and difficult laryngoscopy and tracheal intubation.

B. Measurements We will record morphometric characteristics of all patients. The quality of the airway will be evaluated using the Mallampati, thyromental distance, interincisor gap distance, neck mobility and circumference, and sternomental distance. All intubators will note their laryngoscopy experience level (Cormack-Lehane Scale modified by Yentis, POGO score). Additionally, the anesthesiologist will provide a personal, subjective opinion of a possible difficult laryngoscopy and intubation based on scale from 1 to 5. Any evidence of fogging on the lens will be noted.

Intubation: We will measure the time and number of attempts required for successful endotracheal intubation, easiness of double view (direct vs video), laryngoscopy view change, and any alternative aid (bougie, stylet, etc) required. An attempt is defined as placement of an ETT through the glottic opening and into the trachea. Removal/reinsertion of the laryngoscope or the switching of the laryngoscopist will constitute as a new attempt. Once an optimal positional has been confirmed, position of the ETT will not be further altered. A four question survey will be presented to the resident (is it easy to be used, is it intuitive, do you think it is valuable as a teaching tool, what do you think is the greatest/ worst value of this device).

Degree of irritation: Following intubation in either group, the appearance of oropharynx, pharynx, epiglottis, and arytenoids will be checked. The presence of abrasions, bleeding, redness, perforation or other signs of tissue or dental injury will be recorded.

SUBJECTS:

The subjects will be adult surgical candidates age 18-80, ASA I- III, presenting for elective surgery who require general anesthesia. Patients will be chosen if it is determined that endotracheal intubation is required. Patients will be excluded if they are considered so difficult (i.e. Mallampatti IV, < 2 FB or 4 cm mouth opening), that an awake fiberoptic intubation should be performed. ASA IV and V patients will also be excluded from the study in addition to those who need rapid sequence (i.e. patients with acid reflux) and have known cardiovascular disease

RECRUITMENT METHODS/ INFORMED CONSENT:

Physician investigators will interview all potential subjects to determine if subjects are suitable for the study. Written consent will be obtained by an anesthesiology resident or research assistant.

PROCEDURES TO MAINTAIN CONFIDENTIALITY:

All information recorded on the anesthetic records will be kept strictly confidential and all data will be kept in a data logbook locked in the office of the principal investigator. We will record patients only by study code number.

DATA ANALYSIS:

Data will be analyzed using t- tests, ANOVA, or Fisher Exact test, as appropriate. Results will be presented as means ± SD. P < 0.05 will be considered as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 80 years of age
* ASA I - III
* Mallampati I-III
* Mouthopening > 4cm

Exclusion Criteria:

* Age < 18 years and > 80 years of age
* ASA IV - V
* Mallampati IV - V
* Mouthopening < 4cm

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-02; Primary Completion 2010-09 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Davide Cattano, MD, PhD, Principal Investigator — University of Texas Medical School at Houston
Locations (1):
- Memorial Hermann Hospital, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- C-MAC Direct Laryngoscopy, Then C-MAC Indirect Laryngoscopy; C-MAC Indirect Laryngoscopy, Then C-MAC Direct Laryngoscopy: Each patient received both direct laryngoscopy and indirect laryngoscopy, and the order of receipt was randomized. Patients were intubated once, and intubation occurred after the second laryngoscopy.
Period: Overall Study
Arm/Group | C-MAC Direct Laryngoscopy, Then C-MAC Indirect Laryngoscopy | C-MAC Indirect Laryngoscopy, Then C-MAC Direct Laryngoscopy
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | C-MAC Direct Laryngoscopy, Then C-MAC Indirect Laryngoscopy | C-MAC Indirect Laryngoscopy, Then C-MAC Direct Laryngoscopy | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.2 (14.2) | 49.1 (15.2) | 47.7 (14.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 17 | 35
  Male | 7 | 8 | 15
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Time for Intubation
Description: Time taken for successful placement of endotracheal tube (that is, intubation).
Time Frame: at the time of intubation (about 10 seconds)
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | C-MAC Direct Laryngoscopy, Then C-MAC Indirect Laryngoscopy | C-MAC Indirect Laryngoscopy, Then C-MAC Direct Laryngoscopy
Number analyzed (Participants) | 25 | 25
seconds | 12.3 (11.1) | 9.8 (7.1)

2. Secondary Outcome: Laryngoscopy Time
Description: Laryngoscopy time is defined as the time between advancing the laryngoscopy and obtaining the optimal view of the airway.
Time Frame: at the time of laryngoscopy (about 10 seconds)
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | C-MAC Direct Laryngoscopy, Then C-MAC Indirect Laryngoscopy | C-MAC Indirect Laryngoscopy, Then C-MAC Direct Laryngoscopy
Number analyzed (Participants) | 25 | 25
seconds
  first laryngoscopy | 8.7 (4.7) | 14.1 (12.1)
  second laryngoscopy | 9.1 (6.1) | 12.2 (7.5)

3. Secondary Outcome: Airway View at the Time of Laryngoscopy as Categorized by the Modified Cormack-Lehane Classification (Before External Manipulation)
Description: Modified Cormack-Lehane classification:
  1. Full view of glottis
  2. a Partial view of glottis
  2b Only posterior extremity of glottis seen or only arytenoid cartilages 3 Only epiglottis seen, none of glottis seen 4 Neither glottis nor epiglottis seen
Time Frame: at the time of laryngoscopy (about 10 seconds)
Measure: Count of Participants; unit: Participants
Arm/Group | C-MAC Direct Laryngoscopy, Then C-MAC Indirect Laryngoscopy | C-MAC Indirect Laryngoscopy, Then C-MAC Direct Laryngoscopy
Number analyzed (Participants) | 25 | 25
Participants
  first laryngoscopy: 1 | 12 | 19
  first laryngoscopy: 2a | 7 | 3
  first laryngoscopy: 2b | 6 | 1
  first laryngoscopy: 3 | 0 | 2
  first laryngoscopy: 4 | 0 | 0
  second laryngoscopy: 1 | 20 | 11
  second laryngoscopy: 2a | 4 | 6
  second laryngoscopy: 2b | 1 | 5
  second laryngoscopy: 3 | 0 | 3
  second laryngoscopy: 4 | 0 | 0

4. Secondary Outcome: Airway View at the Time of Laryngoscopy as Categorized by the Modified Cormack-Lehane Classification (After External Manipulation)
Description: as for outcome 3
Time Frame: at the time of laryngoscopy (about 10 seconds)
Measure: Count of Participants; unit: Participants
Arm/Group | C-MAC Direct Laryngoscopy, Then C-MAC Indirect Laryngoscopy | C-MAC Indirect Laryngoscopy, Then C-MAC Direct Laryngoscopy
Number analyzed (Participants) | 25 | 25
Participants
  first laryngoscopy: 1 | 15 | 20
  first laryngoscopy: 2a | 10 | 4
  first laryngoscopy: 2b | 0 | 1
  first laryngoscopy: 3 | 0 | 0
  first laryngoscopy: 4 | 0 | 0
  second laryngoscopy: 1 | 22 | 12
  second laryngoscopy: 2a | 3 | 11
  second laryngoscopy: 2b | 0 | 2
  second laryngoscopy: 3 | 0 | 0
  second laryngoscopy: 4 | 0 | 0

5. Secondary Outcome: Number of Participants With Successful Intubation
Time Frame: at the time of intubation (about 10 seconds)
Measure: Count of Participants; unit: Participants
Arm/Group | C-MAC Direct Laryngoscopy, Then C-MAC Indirect Laryngoscopy | C-MAC Indirect Laryngoscopy, Then C-MAC Direct Laryngoscopy
Number analyzed (Participants) | 25 | 25
Participants | 25 | 25

6. Secondary Outcome: Ease of Intubation as Assessed by a Rating Scale
Description: Ease of intubation as assessed by a rating scale, which ranged from 1 (very easy) to 5 (very difficult).
Time Frame: at the time of intubation (about 10 seconds)
Measure: Count of Participants; unit: Participants
Arm/Group | C-MAC Direct Laryngoscopy, Then C-MAC Indirect Laryngoscopy | C-MAC Indirect Laryngoscopy, Then C-MAC Direct Laryngoscopy
Number analyzed (Participants) | 25 | 25
Participants
  1 | 14 | 16
  2 | 6 | 4
  3 | 4 | 4
  4 | 1 | 1
  5 | 0 | 0

7. Secondary Outcome: Ease of Laryngoscopy as Assessed by a Rating Scale
Description: Ease of laryngoscopy as assessed by a rating scale, which ranged from 1 (very easy) to 5 (very difficult).
Time Frame: at the time of laryngoscopy (about 10 seconds)
Measure: Count of Participants; unit: Participants
Arm/Group | C-MAC Direct Laryngoscopy, Then C-MAC Indirect Laryngoscopy | C-MAC Indirect Laryngoscopy, Then C-MAC Direct Laryngoscopy
Number analyzed (Participants) | 25 | 25
Participants
  1 | 15 | 13
  2 | 5 | 4
  3 | 4 | 5
  4 | 1 | 3
  5 | 0 | 0

ADVERSE EVENTS:
Time Frame: About 2 hours
Arm/Group | C-MAC Direct Laryngoscopy, Then C-MAC Indirect Laryngoscopy | C-MAC Indirect Laryngoscopy, Then C-MAC Direct Laryngoscopy
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes